CLINICAL TRIAL: NCT02741310
Title: Phase 1, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Effect on Blood Pressure of AMG 334 Given Concomitantly With Subcutaneous Sumatriptan (Imitrex™) in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Erenumab on Blood Pressure When Given Concomitantly With Subcutaneous Sumatriptan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140255; 2015-004537-28 (EudraCT Number)
Record Dates: First submitted 2016-02-19; First posted 2016-04-18 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Sumatriptan; erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received a placebo intravenous (IV) infusion on day 1 then 12 mg subcutaneous sumatriptan on day 2 (Part 1). After a 2-day washout participants received another placebo IV infusion on day 4 followed by 12 mg subcutaneous sumatriptan on day 5 (Part 2).
  Interventions: Drug: Placebo; Drug: Sumatriptan
- Erenumab (Experimental): Participants received a placebo intravenous (IV) infusion on day 1 then 12 mg subcutaneous sumatriptan on day 2 (Part 1). After a 2-day washout participants received 140 mg erenumab IV infusion on day 4 followed by 12 mg subcutaneous sumatriptan on day 5 (Part 2).
  Interventions: Drug: Placebo; Drug: Sumatriptan; Drug: Erenumab

INTERVENTIONS:
Drug: Placebo — Administered by intravenous infusion
Drug: Sumatriptan — Administered by two 6 mg subcutaneous injections 1 hour apart on day 2 and day 5
  Other Names: Imitrex™
Drug: Erenumab — Administered by intravenous infusion
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab

SUMMARY:
The primary objective of this study was to assess the effects of subcutaneous sumatriptan alone and the effects of a single dose of erenumab (AMG 334) intravenous (IV) and sumatriptan concomitant therapy on resting blood pressure in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects ≥ 18 to ≤ 55 years old
* Good general health
* Laboratory results within range
* Other Inclusion Criteria May Apply

Exclusion Criteria:

* Female subjects pregnant or breastfeeding
* An unstable medical condition
* History of cancer
* Active liver disease
* Positive Hepatitis B or Hepatitis C
* Unwilling or unable to limit alcohol consumption
* Unable to refrain from strenuous exercise
* Other Exclusion Criteria May Apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Leuven, Belgium

REFERENCES:
- [Background] de Hoon J, Van Hecken A, Vandermeulen C, Herbots M, Kubo Y, Lee E, Eisele O, Vargas G, Gabriel K. Phase 1, randomized, parallel-group, double-blind, placebo-controlled trial to evaluate the effects of erenumab (AMG 334) and concomitant sumatriptan on blood pressure in healthy volunteers. Cephalalgia. 2019 Jan;39(1):100-110. doi: 10.1177/0333102418776017. Epub 2018 May 21. PMID 29783863
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 center in Belgium; participants were enrolled from 22 February 2016 to 11 May 2016.
Pre-assignment Details: Eligible participants were randomized on day 1 to receive either erenumab or matching placebo in a 2:1 allocation ratio.
Groups:
- Group A: Placebo + Sumatriptan: Participants received a placebo intravenous (IV) infusion on day 1 then 12 mg subcutaneous (SC) sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 2 (Part 1). After a 2-day washout participants received another placebo IV infusion on day 4 followed by 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 5 (Part 2).
- Group B: Erenumab + Sumatriptan: Participants received a placebo IV infusion on day 1 then 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 2 (Part 1). After a 2-day washout participants received 140 mg erenumab IV infusion on day 4 followed by 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 5 (Part 2).
Period: Overall Study
Arm/Group | Group A: Placebo + Sumatriptan | Group B: Erenumab + Sumatriptan
Started | 12 | 22
Completed | 10 | 20
Not Completed | 2 | 2
Not completed — Sponsor Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Placebo + Sumatriptan | Group B: Erenumab + Sumatriptan | Total
Number analyzed (Participants) | 12 | 22 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (8.6) | 29.1 (10.3) | 28.5 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  18 - 24 years | 6 | 9 | 15
  25 - 55 years | 6 | 13 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 16 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 22 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black (or African American) | 0 | 1 | 1
  Multiple | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 12 | 21 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Averages of Mean Arterial Pressure
Description: Mean arterial pressure (MAP) is the average arterial pressure during a single cardiac cycle. MAP was calculated as diastolic blood pressure (DBP) + 0.33 * (systolic blood pressure [SBP]-DBP). Individual time-weighted average in MAP were calculated as area under the measurement-time curve from predose through 2.5 hours of MAP divided by the time period over which the measurements were made (ie, AUCmap0-2.5 hr /2.5 hours).
  Data were analyzed using a linear mixed effects regression model with fixed effects for treatment and period and random effect for subject; Sumatriptan Alone data include participants from both Groups A (Parts 1 and 2) and B (Part 1 only).
Time Frame: Days 2 and 5 from predose to 2.5 hours after sumatriptan dosing.
Population: All participants who received at least 1 dose of study drug (placebo, sumatriptan, or erenumab) and with available data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Sumatriptan Alone: All participants who received placebo and sumatriptan (Group A, Parts 1 and 2 and Group B, Part 1).
- Erenumab + Sumatriptan: All participants who received erenumab plus sumatriptan (Group B, Part 2)
Arm/Group | Sumatriptan Alone | Erenumab + Sumatriptan
Number analyzed (Participants) | 34 | 20
mmHg | 87.40 (0.98) | 87.36 (1.22)
Statistical Analysis 1: Comparison: Sumatriptan Alone vs Erenumab + Sumatriptan; A linear mixed effects regression analysis was performed to assess if the time-weighted average in MAP for erenumab with sumatriptan is similar to sumatriptan alone. A two-sided 90% confidence interval (equivalent to a one-sided upper 95% CI) for the mean treatment difference was calculated using a linear mixed-effects model with fixed effects for treatment and period and a random effect for subject; Test type: Other — The clinical hypothesis was that there would be no clinically meaningful difference between the blood pressure effects of sumatriptan alone and the effects of a single dose of erenumab IV and sumatriptan concomitant therapy. A clinically meaningful difference was defined as the upper bound of the 90% confidence interval (CI) of treatment difference between erenumab IV and sumatriptan compared to sumatriptan alone being ≥ 5 mmHg on the time-weighted scale resting MAP; LS Mean Difference = -0.04, 90% CI 2-sided [-2.16 to 2.08]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and according to the following:
  Grade 1 = Mild AE, asymptomatic or mild symptoms; Grade 2 = Moderate, minimal, local or noninvasive intervention indicated; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences, urgent intervention indicated; Grade 5 = Death related to AE.
Time Frame: From the first dose of study drug (sumatriptan, placebo or erenumab) until 84 days after the last dose (89 days). Part 1 includes AEs from day 1 to predose on day 4 and Part 2 includes AEs from day 4 through day 89.
Population: All participants who received at least 1 dose of study drug (placebo, sumatriptan, or erenumab).
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Group A: Placebo + Sumatriptan: In Part 1 participants in Group A received a placebo IV infusion on day 1 then 12 mg SC sumatriptan on day 2.
- Part 1 Group B: Placebo + Sumatriptan: In Part 1 participants in Group B received a placebo IV infusion on day 1 then 12 mg SC sumatriptan on day 2.
- Part 2 Group A: Placebo + Sumatriptan: In Part 2 participants in Group A received another placebo IV infusion on day 4 followed by 12 mg SC sumatriptan on day 5.
- Part 2 Group B: Erenumab + Sumatriptan: In Part 2 participants in Group B received 140 mg erenumab IV infusion on day 4 followed by 12 mg SC sumatriptan on day 5.
Arm/Group | Part 1 Group A: Placebo + Sumatriptan | Part 1 Group B: Placebo + Sumatriptan | Part 2 Group A: Placebo + Sumatriptan | Part 2 Group B: Erenumab + Sumatriptan
Number analyzed (Participants) | 12 | 22 | 12 | 22
Participants
  Any adverse event | 11 | 19 | 9 | 17
  Adverse event ≥ grade 2 | 1 | 0 | 0 | 3
  Adverse event ≥ grade 3 | 0 | 0 | 0 | 0
  Adverse event ≥ grade 4 | 0 | 0 | 0 | 0
  Serious adverse events | 0 | 0 | 0 | 0
  AE leading to discontinuation of study drug | 2 | 2 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0

3. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 6 Hours for Sumatriptan
Description: Plasma concentrations of sumatriptan were quantified using a validated high performance liquid chromatographic method with tandem mass spectrometry detection.
  Area under the plasma concentration-time curve from time 0 to 6 hours post dose (AUC6hr) after the 2nd 6 mg dose of sumatriptan was estimated using the linear trapezoidal method. Sumatriptan plasma concentrations below the lower limit of quantification (LLOQ; 0.100 ng/mL) were set to 0 before data analysis.
  Log-transformed AUC6hr was analyzed using a linear mixed effects model with treatment as a fixed effect and subject as a random effect.
  Sumatriptan Alone data include participants from both Groups A (Parts 1 and 2) and B (Part 1 only).
Time Frame: Day 2 and day 5 at 1 hour (prior to 2nd sumatriptan injection), 1 hour 10 minutes, 1.25, 1.5, 2, 3, 4.5, and 7 hours relative to the first 6 mg dose of sumatriptan.
Population: All participants who received at least 1 dose of study drug (placebo, sumatriptan, or erenumab) and have at least one pharmacokinetic (PK) sample collected or one PK parameter.
Measure: Geometric Least Squares Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Sumatriptan Alone | Erenumab + Sumatriptan
Number analyzed (Participants) | 30 | 20
hr*ng/mL | 133.33 (1.03) | 130.59 (1.04)
Statistical Analysis 1: Comparison: Sumatriptan Alone vs Erenumab + Sumatriptan; The mean for each treatment was compared using a linear mixed effects model with group A (sumatriptan alone) as the reference treatment group. The linear mixed effects model included treatment (erenumab with sumatriptan vs sumatriptan alone) and period as a fixed effect and subject as a random effect; Test type: Other; Geometric Least Squares Mean Ratio = 0.98, 90% CI 2-sided [0.93 to 1.03]

4. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity for Sumatriptan
Description: Plasma concentrations of sumatriptan were quantified using a validated high performance liquid chromatographic method with tandem mass spectrometry detection. The area under the plasma concentration-time curve from time 0 to infinity (AUCinf) after the 2nd 6 mg dose of sumatriptan was estimated as the sum of AUClast and Clast/λz where Clast is the last observed concentration and λz is the first-order terminal rate constant estimated via linear regression of the terminal log-linear decay phase. Sumatriptan plasma concentrations below the lower limit of quantification (LLOQ) (0.100 ng/mL) were set to 0 before data analysis.
  Log-transformed AUCinf was analyzed using a linear mixed effects model with treatment as a fixed effect and subject as a random effect. Sumatriptan Alone data include participants from both Groups A (Parts 1 and 2) and B (Part 1 only).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Sumatriptan Alone | Erenumab + Sumatriptan
Number analyzed (Participants) | 30 | 20
hr*ng/mL | 144.32 (1.03) | 144.81 (1.04)
Statistical Analysis 1: Comparison: Sumatriptan Alone vs Erenumab + Sumatriptan; [analysis description as in outcome 3, analysis 1]; Test type: Other; Geometric Least Squares Mean Ratio = 1.00, 90% CI 2-sided [0.96 to 1.05]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sumatriptan
Description: Plasma concentrations of sumatriptan were quantified using a validated high performance liquid chromatographic method with tandem mass spectrometry detection. Sumatriptan plasma concentrations below the lower limit of quantification (LLOQ) (0.100 ng/mL) were set to 0 before data analysis.
  Log-transformed maximum observed plasma concentration (Cmax) was analyzed using a linear mixed effects model with treatment as a fixed effect and subject as a random effect. Sumatriptan Alone data include participants from both Groups A (Parts 1 and 2) and B (Part 1 only).
Time Frame: Day 2 and day 5 at predose, 1 hour (prior to 2nd sumatriptan injection), 1 hour 10 minutes, 1.25, 1.5, 2, 3, 4.5, and 7 hours relative to the first 6 mg dose of sumatriptan.
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Sumatriptan Alone | Erenumab + Sumatriptan
Number analyzed (Participants) | 30 | 20
ng/mL | 83.50 (1.05) | 79.00 (1.07)
Statistical Analysis 1: Comparison: Sumatriptan Alone vs Erenumab + Sumatriptan; [analysis description as in outcome 3, analysis 1]; Test type: Other; Geometric Least Squares Mean Ratio = 0.95, 90% CI 2-sided [0.82 to 1.09]

6. Secondary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies
Description: Two validated assays were used to detect the presence of anti-erenumab antibodies. All samples were first tested in an electrochemiluminescence-based bridging assay to detect antibodies capable of binding to erenumab (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based assay to determine neutralizing activity against erenumab (Neutralizing Antibody Assay). If a post-dose sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
  Binding/neutralizing antibody positive is defined as participants with an antibody positive postbaseline results and with a negative or no result at baseline.
Time Frame: Baseline and day 89
Population: Participants who received at least 1 dose of study drug (placebo, sumatriptan, or erenumab) with a postbaseline antibody result.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Placebo + Sumatriptan | Group B: Erenumab + Sumatriptan
Number analyzed (Participants) | 10 | 20
Participants
  Binding antibody positive | 0 | 1
  Neutralizing antibody positive | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (sumatriptan, placebo or erenumab) until 84 days after the last dose (89 days). Part 1 includes AEs from day 1 to predose on day 4 and Part 2 includes AEs from day 4 through day 89.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Part 1 Group A: Placebo + Sumatriptan: In Part 1 participants in Group A received a placebo IV infusion on day 1 then 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 2.
- Part 1 Group B: Placebo + Sumatriptan: In Part 1 participants in Group B received a placebo IV infusion on day 1 then 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 2.
- Part 2 Group A: Placebo + Sumatriptan: In Part 2 participants in Group A received another placebo IV infusion on day 4 followed by 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 5.
- Part 2: Group B: Erenumab + Sumatriptan: In part 2 participants in Group B received 140 mg erenumab IV infusion on day 4 followed by 12 mg SC sumatriptan (6 mg, followed by 6 mg at least 1 hour later) on day 5.
Arm/Group | Part 1 Group A: Placebo + Sumatriptan | Part 1 Group B: Placebo + Sumatriptan | Part 2 Group A: Placebo + Sumatriptan | Part 2: Group B: Erenumab + Sumatriptan
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/22 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 11/12 | 17/22 | 9/10 | 17/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Group A: Placebo + Sumatriptan (N=12) | Part 1 Group B: Placebo + Sumatriptan (N=22) | Part 2 Group A: Placebo + Sumatriptan (N=10) | Part 2: Group B: Erenumab + Sumatriptan (N=20)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Discomfort (General disorders) | 4 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 1 | 1 | 1 | 1
Injection site erythema (General disorders) | 2 | 4 | 1 | 2
Injection site swelling (General disorders) | 2 | 4 | 1 | 2
Injection site urticaria (General disorders) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 1 | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4
Burning sensation (Nervous system disorders) | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1
Head discomfort (Nervous system disorders) | 4 | 8 | 3 | 8
Headache (Nervous system disorders) | 1 | 3 | 0 | 4
Paraesthesia (Nervous system disorders) | 4 | 3 | 4 | 4
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 3
Leukocyturia (Renal and urinary disorders) | 1 | 1 | 0 | 1
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.